CLINICAL TRIAL: NCT01143207
Title: Pharmacokinetics of Subcutaneous Depot Medroxyprogesterone Acetate Injected in the Upper Arm
Brief Title: PK of Depo SubQ Injected in the Upper Arm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10206
Record Dates: First submitted 2010-06-07; First posted 2010-06-14 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Contraception
Keywords: AE adverse event; DCF data collection forms; DMC Data Monitoring Committee; FDA U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; ICH International Conference of Harmonisation; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); SAE serious adverse event; µg microgram; ULN upper limit of the normal range
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medroxyprogesterone acetate (Experimental): Single injection of Medroxyprogesterone acetate (hormonal contraceptive)
  Interventions: Drug: Medroxyprogesterone acetate

INTERVENTIONS:
Drug: Medroxyprogesterone acetate — Injectable hormonal contraceptive
  Other Names: Depo-SubQ Provera 104

SUMMARY:
A single-arm trial to demonstrate that Depo-SubQ Provera injected in the upper arm is adequate for effective contraception

DETAILED DESCRIPTION:
A single-arm trial to demonstrate that the blood levels of medroxyprogesterone acetate are adequate for effective contraception when Depo-SubQ Provera 104 is injected in the upper arm

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40
* negative pregnancy test on day of injection
* not wishing to become pregnant in the next 12 months
* at negligible risk of pregnancy (e.g. sterilized, in exclusively same-gender partnership, in a monogamous relationship with vasectomized partner, abstinent, using non-hormonal IUD)
* body mass index of 18-30

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Archer, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Clinical Research Center, Dept. of Obstetrics & Gynegology, Eastern Virginia Medical School, Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medroxyprogesterone Acetate: Single injection of Medroxyprogesterone acetate (hormonal contraceptive)
  Medroxyprogesterone acetate : Injectable hormonal contraceptive
Period: Overall Study
Arm/Group | Medroxyprogesterone Acetate
Started | 26
Completed | 24
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximal Serum Concentration of Medroxyprogesterone Acetate (MPA))
Time Frame: 120 days following injection
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 25
ng/mL | 0.953 (0.308) [2 to 14]

2. Primary Outcome: Tmax (Time to Cmax)
Time Frame: 120 days following injection
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 25
days | 8 [2 to 14]

3. Primary Outcome: AUC 0-91 (Area Under Curve)
Time Frame: first 91 days following injection
Measure: Mean (Standard Deviation); unit: ng day/mL
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 24
ng day/mL | 45.1 (14.5)

4. Primary Outcome: MPA Concentration at Day 91 (C91)
Time Frame: day 91 after first injection
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 22
ng/mL | 0.427 (0.354)

5. Primary Outcome: MPA Concentration at Day 104 (C104)
Time Frame: day 104 after injection
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 23
ng/mL | 0.366 (0.278)

6. Primary Outcome: MPA Concentration at Day 120 (C120)
Time Frame: day 120 after injection
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Medroxyprogesterone Acetate
Number analyzed (Participants) | 23
ng/mL | 0.327 (0.206)

ADVERSE EVENTS:
Arm/Group | Medroxyprogesterone Acetate
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medroxyprogesterone Acetate (N=26)
Bipolar Disorder (Psychiatric disorders) | 1 (1) — exacerbation of pre-existing Bipolar Disorder
Hysterectomy (Surgical and medical procedures) | 1 (1) — total abdominal hysterectomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medroxyprogesterone Acetate (N=26)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
vaginal infection (bacterial vaginosis) (Reproductive system and breast disorders) | 2 (2)
bladder pain (Renal and urinary disorders) | 1 (1)
Biopsy breast (Investigations) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dental infection (Infections and infestations) | 1 (1)
Dental pain (Gastrointestinal disorders) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dispepsia (Gastrointestinal disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Corneal abrasion (Eye disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (sinus congestion) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (sinus headache) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Vulvovaginal candidiasis (yeast infection) (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal candidiasis (vaginal yeast infection) (Reproductive system and breast disorders) | 1 (1)
sinusitis (congestion) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No